CLINICAL TRIAL: NCT04905836
Title: Treatment of COVID-19-Induced Acute Respiratory Distress: A Phase 2 Study of Intravenous Administration of Allogeneic Adipose-Derived Mesenchymal Stem Cells
Brief Title: Study of Allogeneic Adipose-Derived Mesenchymal Stem Cells for Treatment of COVID-19 Acute Respiratory Distress
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-COV-202
Record Dates: First submitted 2021-05-27; First posted 2021-05-28 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-MSC (Experimental): Subjects will receive intravenous infusions of COVI-MSC (two vials or a total of ≈ 30 million cells) on Day 0, Day 2, and Day 4
  Interventions: Biological: COVI-MSC
- Placebo (Placebo Comparator): Subjects will receive intravenous infusions of placebo (two vials) on Day 0, Day 2, and Day 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-MSC — COVI-MSC are allogeneic culture-expanded adipose-derived mesenchymal stem cells
  Arms: COVI-MSC
Drug: Placebo — Excipient solution
  Arms: Placebo

SUMMARY:
This is a Phase 2 study to assess COVI-MSC in the setting of current standard of care in hospitalized subjects with RT-PCR confirmed SARS-CoV-2 (COVID-19) infection and acute respiratory distress / acute respiratory distress syndrome.

DETAILED DESCRIPTION:
This is a Phase 2 multicenter (United States and Mexico) study to assess the safety and preliminary efficacy of COVI-MSC in the setting of current standard of care in hospitalized subjects with RT-PCR confirmed SARS-CoV-2 (COVID-19) infection and acute respiratory stress (ARD) / acute respiratory distress syndrome (ARDS).

Subjects will be randomized 1:1 COVI-MSC to placebo. COVI-MSC or placebo will be administered intravenously on Day 0, Day 2, and Day 4.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed SARS-CoV-2 infection as determined by an approved polymerase chain reaction (PCR) or an approved antigen test of any specimen (can be documented from inpatient medical record)
* Hospitalized with at least "severe" COVID-19-induced ARD or ARDS as defined per FDA Guidance; COVID-19: Developing Drugs and Biological Products for Treatment or Prevention
* Requires oxygen supplementation at Screening
* Willing to follow contraception guidelines

Exclusion Criteria:

* Current standard of care treatments for COVID-19 appear to be working and the subject is clinically improving
* Has severe ARDS with a PaO2/FiO2 (PF ratio) ≤ 100 mmHg or SpO2/FiO2 ratio < 150 mmHg with PEEP ≥ 5cm H2O
* A previous stem cell infusion unrelated to this trial
* Pregnant or breast feeding or planning for either during the study
* Suspected uncontrolled active bacterial, fungal, viral, or other infection (aside from infection with COVID-19)
* History of a splenectomy, lung transplant or lung lobectomy
* Concurrent participation in another clinical trial involving therapeutic interventions (observational study participation is acceptable)
* Expected survival or time to withdrawal of life-sustaining treatments expected to be < 7 days
* Has an existing "Do Not Intubate" order
* Has undergone home mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure (CPAP/BIPAP) used solely for sleep-disordered breathing (eg, obstructive sleep apnea)
* Has any significant medical condition, laboratory abnormality or psychiatric illness that in the investigator's opinion would interfere or prevent the subject from safely participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate at Day 28 | Baseline through Day 28
  All-cause mortality rate at Day 28
Incidence of all adverse events (AEs) (safety) | Baseline through study completion at Day 90
  Safety as assessed by incidence of AEs by type, frequency, severity, and causality using the Common Terminology Criteria for Adverse Events, Version 5 (CTCAEv5)
Incidence of treatment-emergent adverse events (safety) | Baseline through study completion at Day 90
  Safety as assessed by incidence of treatment-emergent AEs (TEAEs) by type, frequency, severity, and causality using CTCAEv5 criteria
Incidence of severe adverse events (safety) | Baseline through study completion at Day 90
  Safety as assessed by incidence of serious AEs (SAEs) by type, frequency, severity, and causality using CTCAEv5 criteria
Incidence of infusion-related adverse events (safety) | Baseline to Hour 4
  Safety as assessed by incidence of Infusion-related AEs (IrAEs) by type, frequency, severity, and causality using CTCAEv5 criteria over 4 hours

SECONDARY OUTCOMES:
All-cause mortality rate at Day 60 and 90 | Baseline through Day 60 and Day 90
  All-cause mortality rate at Day 60 and 90
Number of ventilator-free days through Day 28 | Baseline through Day 28
  Number of ventilator-free days through Day 28
Number of ICU days through Day 28 | Baseline through Day 28
  Number of ICU days through day 28
Change in clinical status | Baseline to Day 28
  Change in clinical status as assessed using the WHO Clinical Progression Scale (0-10 scale, where lower score means a better outcome) at Day 28
Change in oxygenation | Baseline to Day 14 Day 28, and Day 60
  Change in oxygenation as assessed using PaO2:FiO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (6):
- United States (6):
  - Teradan Clinical Trials LLC, Brandon, Florida
  - Sarasota Memorial Health Care System (SMH), Sarasota, Florida
  - St Luke's Research, Boise, Idaho
  - St. Luke's Boise, Boise, Idaho
  - Ascension St. John, Tulsa, Oklahoma
  - PRX Research/Dallas Regional Medical Center, Mesquite, Texas